CLINICAL TRIAL: NCT02487641
Title: Obese Pregnant Women: Optimizing Mid-trimester Fetal Ultrasound for Risk Estimation During Pregnancy and Childhood
Brief Title: Obese Pregnant Women: Optimizing Fetal Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Holbaek Sygehus (Other)
Collaborators: Odense University Hospital (Other); Technical University of Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: 12-000095
Record Dates: First submitted 2015-06-23; First posted 2015-07-01 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Obesity; Fetal Malformation
Keywords: Ultrasound; mid-trimester; Obesity; pregnancy
MeSH Terms: conditions — Obesity; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Moderat Obesity: 60 persons with BMI between 30-34.49 kg/m2
- Sever Obesity: 60 persons with BMI above 34.49 kg/m2
- Normal weighted: 60 persons with BMI between 18.5-24.49 kg/m2

SUMMARY:
This study aim to evaluate the quality of fetal ultrasound in obese pregnant women. The hypotheses is that an early ultrasound will improve the quality of the ultrasound in obese.

DETAILED DESCRIPTION:
Ultrasound examination for fetal anomaly is especially challenging in obese gravida. The foetus is more likely to have congenital anomalies and imaging in these patients is technically more difficult.

The investigators hypotheses that an earlier ultrasound with alternative technics will improve the quality and thereby improve the identification of anomalies. By using transvaginal ultrasound and abdominal ultrasound at the window just above the symphysis, were the subcutaneous fat is known to be thinner, the investigators hope to achieve a better overview. This will be done by evaluating fetal ultrasound at three different gestational ages (GA); GA 13, 15 and 21 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* BMI ≥ 30 Kg/m2
* BMI: 18,5-25 Kg/m2
* Understand and speak Danish and thereby be able to give confirmed consent.

Exclusion Criteria:

* Multiple gestations
* Overweight (BMI: 25-29,9 Kg/m2)
* Alcohol or drug abuse
* Chronically diseases before pregnancy as diabetes, hypertension, or thyroid diseases
* Gastric bypass or other obesity related surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sixty pregnant women with BMI ≥ 30 Kg/m2, 60 pregnant women with BMI ≥ 35 Kg/m2 and 60 Kg/m2 pregnant women normal weighted (BMI: 18,5-24,9 Kg/m2) will be included.
  Women will be classified by their pre-pregnancy BMI and all pregnant women with an age ≥ 18 will be offered to attend the project and those who accept will be admitted. The recruitment will be performed at Holbæk Hospital and Odense University Hospital.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Image quality of ultrasound at 15 compared with 21 weeks of gestation. | The participants will be examined for an hour at to different stages of the pregnancy (GA 14+0-15+0, GA 20+0-21+0)
  Image quality evaluated by experts on a visual analog scale from +50 - -50, parried with standardized ultrasound pictures at the above mentioned GA.

SECONDARY OUTCOMES:
Image quality of ultrasound at 13 compared with 15 weeks of gestation. | The participants will be examined for an hour at to different stages of the pregnancy (GA 11+3 - 13+0, GA 14+0-15+0)
  Image quality evaluated by experts on a visual analog scale from +50 - -50, parried with standardized ultrasound pictures at the above mentioned GA.
Analyses of BMI, visceral to subcutaneous fat ratio, distance from cutis to amnion and hip-waist ratio´s influence on image quality. | The participants will be examined for an hour at three different stages of the pregnancy (GA 13, GA 15, GA 21 and GA 36 weeks).
Weight estimate | The participants will be examined for an hour at GA 36 weeks. The participants will in all be followed until 6 months after birth, which is one year in all.
  The use of weight estimate in obese pregnant women at GA 36 compared to birthweight.
Amnion fluid in obese | The participants will be examined for an hour at three different stages of the pregnancy (GA 15, GA 21, GA 36 weeks)
  Measurement of amnion fluid by deepest vertical pocket and amnion fluid index.
Crown-rump length (CRL) measurement transvaginal and abdominal | The participants will be examined for an hour at GA 13 weeks.
  Measurement of CRL in mm, by using two different probes, transvaginal and abdominal.

CONTACTS AND LOCATIONS:
Overall Officials: Ida Näslund Thagaard, M.D., Principal Investigator — Department of obstetrics and gynecology, Holbæk Hospital, Denmark
Locations (1):
- Department of Gynaechology and Obstetrics, Holbaek Hospital, Holbæk, Denmark